CLINICAL TRIAL: NCT05642793
Title: Effect of Postvitrectomy Proactive Use of Conbercept on Postoperative Complications in PDR Patients
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Peking University Third Hospital (Other)
Responsible Party: Principal Investigator, Chen Huijin, Clinical Professor, Peking University Third Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: PDR vitrectomy1
Record Dates: First submitted 2022-11-30; First posted 2022-12-08 (Actual); Last update posted 2022-12-14 (Actual); Status verified 2022-12

CONDITIONS: Proliferative Diabetic Retinopathy
Keywords: vitrectomy
MeSH Terms: interventions — KH902 fusion protein

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- group 1 (proactive use of conbercept after vitrectomy) (Experimental): proactive use of conbercept after vitrectomy
  Interventions: Drug: proactive Anti-VEGF (conbercept) use
- group 2 (passive use of conbercept after vitrectomy) (Experimental): passive use of conbercept after vitrectomy
  Interventions: Drug: passive Anti-VEGF (conbercept) use

INTERVENTIONS:
Drug: proactive Anti-VEGF (conbercept) use — preventive intravitreal injection of conbercept 2 weeks after vitrectomy, and repeat at 5 weeks and 8 weeks if either of the following is present: intravitreal VEGF concentration at 2 weeks postop is higher than 100 pg/ml, or clinical presentation of DME, VH or NVG.
  Arms: group 1 (proactive use of conbercept after vitrectomy)
Drug: passive Anti-VEGF (conbercept) use — No intravitreal injection of conbercept is used until the patient present with postoperative DME, VH, NVG
  Arms: group 2 (passive use of conbercept after vitrectomy)

SUMMARY:
This is an unmasking randomized clinical trial. the main purpose of this study is to analyze whether posvitrectomy proactive use of conbercept can reduce the rate of postoperative complication in PDR patients.

ELIGIBILITY:
Inclusion Criteria:

* PDR patients undergoing vitrectomy

Exclusion Criteria:

* patients who had received intravitreal injection or systemic use of all types of anti-VEGF agents in the recent three months before vitrectomy
* patients who had received intravitreal injection or systemic use of all types of steroid in the recent one month before vitrectomy
* patients who had received complete PRP before vitrectomy
* patients who are pregnant

Ages: 19 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2022-04-01 (Actual); Primary Completion 2023-09-30 (Estimated); Study Completion 2024-03-01 (Estimated)

PRIMARY OUTCOMES:
rate of postvitrectomy complication | 6 months
  postvitrectomy DME, VH (recurrent or nonabsorbent), NVG

SECONDARY OUTCOMES:
postvitrectomy BCVA | 6 months
  BCVA at 1,3,6 month after vitrectomy

CONTACTS AND LOCATIONS:
Overall Officials: Huijin Chen, Dr., Principal Investigator — Peking University Third Hospital
Locations (1):
- Peking University Third Hospital, Beijing, Beijing Municipality, China